CLINICAL TRIAL: NCT06867770
Title: What is the Proportion of Complications Observed in Infants ≤ 24 Months with a Mild TC (Glasgow ≥ 13) with an Isolated Skull Fracture on the CT Scan (carried Out from H4 of the TC) and Hospitalized At the HFME from 2017 to 2021
Brief Title: Proportion of Complications in Infants with an Isolated Skull Fracture Following Mild TC.
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 878
Record Dates: First submitted 2025-02-24; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Head Trauma; Isolated Skull Fracture; Pediatric; Head Trauma Injury
Keywords: infants; Head trauma; isolated skull fracture; pediatric
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infants aged 24 months or less coming to the emergency department with the discovery of an isolated: * Infant 24 months or less
  * presenting to the pediatric emergencies of HFME
  * for mild head trauma, defined by a Glasgow score greater than or equal to 13,
  * having a scanner at least H4 from their TC
  * and having an isolated skull fracture
  Interventions: Behavioral: Observe the frequency of clinical or paraclinical complications during the hospitalization of these children.

INTERVENTIONS:
Behavioral: Observe the frequency of clinical or paraclinical complications during the hospitalization of these children. — The goal is to collect data on the files of infants hospitalized at the HFME from 2017 to 2021 for monitoring a isolated skull. The data that will be collected are an integral part of the child's care and pre-exist the study. This data will be anonymized and no interaction with the patient is envisaged.

SUMMARY:
Childhood head trauma (TC) is a frequent reason for emergency visits. A bibliographic summary published by Santé Publique France reveals an annual incidence of CD among 0-4 year olds estimated at around 1,340 cases per 100,000 inhabitants in the United States, of which 11% would be intentional (i.e. linked to abuse).

The child presents specificities due to the characteristics of his development, such as :

* the weight of his head, in proportion to his body, is more important compared to the adult;
* the brain is richer in water;
* the bones of the skull are more mouldable and elastic. For these reasons, CD in children has very different consequences from adults, hence the need for a good knowledge of the subject for prevention, management and optimal monitoring of CD in children.

Within the Hospital Femme Mère Enfant (HFME), the procedure consists in hospitalizing all the children presenting a fracture of the skull. They systematically benefit from clinical monitoring, fundoscopy, an electroencephalogram (EEG) and a 3-month consultation with a neurosurgeon to eliminate any complications, but also to detect the inflicted head trauma.

This treatment entails hospitalization for several days for the child and the parents.

The question of the invariability of this local protocol arises because it entails:

* for the parents, linked to the meaning they give to hospitalization
* carrying out several additional examinations for the infant
* a duration of hospitalization which can be extended while waiting for the availability of para-clinical examinations.

Today, HFME specialists intuitively feel that the complication rate is low. In the literature, there are several articles relating the evolution of these children with an isolated fracture of the skull. A review of the literature shows that only 8 out of 5,000 patients had an aggravation of their scanner (such as the appearance of haemorrhage) and none were operated on. Other studies tend to show the absence of deaths, a very low rate of surgery or neurological deficit. There is a suspicion of abuse in 1 to 20% of cases.

Some studies go even further by proposing and evaluating service protocols allowing simple monitoring in the emergency room, then a return home for children with a skull fracture without intracranial lesion and a Glasgow score ≥ 14. These latest studies therefore put general practitioners and paediatricians back in the front line for the follow-up, even in the short term, of infants with an isolated skull fracture.

This study would make it possible to quantify the complications of mild head trauma (Glasgow 13-15) with isolated skull fracture in infants hospitalized in the HFME, and this with unpublished data (electroencephalogram and fundoscopy). According to the results obtained, this could lead to the modification of the care of infants by proposing a reduction in additional examinations and hospitalization, by introducing outpatient monitoring, and this without putting the infant in danger or neglecting inflicted head truama.

ELIGIBILITY:
* Inclusion Criteria * :

  * Infant 24 months or less
  * presenting to the pediatric emergencies of HFME
  * for mild head trauma, defined by a Glasgow score greater than or equal to 13,
  * having a scanner at least H4 from their TC
  * and having an isolated skull fracture
* Exclusion Criteria * :

  * Birth-related trauma
  * history of neurosurgery
  * history of brain tumor
  * Polytrauma
  * Public road accident
  * Personal encephalopathy ATCD
  * Bleeding disorder
  * Anticoagulant treatment
  * Known epilepsy
  * Medium TC and Grace
  * Added presence of hemorrhage, edema or axonal lesion on the initial CT scan

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be taken from children who came to the pediatric emergency room of HFME for a head trauma from January 1, 2017 to December 31, 2021. *
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
frequency of clinical or paraclinical complications during the hospitalization of these children. | - During the hospitalisation - During the consultations organized 3 months after the head trauma.
  * Death
  * Need for surgery
  * - Change in the patient's neurological state: decrease in Glasgow score, convulsion, neurological deficit

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère Enfant, Bron, France